CLINICAL TRIAL: NCT02302716
Title: A Prospective, Randomized, Open-Label Comparison of a Long-Acting Basal Insulin Analog LY2963016 to LANTUS® in Adult Patients With Type 2 Diabetes Mellitus: The ELEMENT 5 Study
Brief Title: A Study of LY2963016 Compared to LANTUS® in Adult Participants With Type 2 Diabetes Mellitus
Acronym: ELEMENT 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15615; I4L-MC-ABER (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 (Experimental): Insulin naive participants started on 10 units (U) LY2963016 given subcutaneously (SC) once a day (QD) for 24 weeks. Participants entering the study on LANTUS®, insulin detemir or neutral protamine hagedorn (NPH) QD will begin the study at their current dose SC. Participants will self titrate LY2963016 based on fasting blood glucose (FBG). Participants entering on insulin detemir or NPH twice a day will be started at 80% of the total daily dose SC. Participants will continue oral antihyperglycemic medication (OAM).
  Interventions: Drug: LY2963016; Drug: Oral Antihyperglycemic Medication
- LANTUS® (Active Comparator): Insulin naive participants started on 10 U LANTUS® given SC QD for 24 weeks. Participants entering the study on LANTUS®, insulin detemir or NPH QD will be started at the same dose SC. Participants entering on insulin detemir or NPH twice a day will be started at 80% of the total daily dose SC. Participants will self titrate LANTUS® based on FBG. Participants will continue OAM.
  Interventions: Drug: LANTUS®; Drug: Oral Antihyperglycemic Medication

INTERVENTIONS:
Drug: LY2963016 — Administered SC
  Arms: LY2963016
Drug: LANTUS® — Administered SC
  Arms: LANTUS®
Drug: Oral Antihyperglycemic Medication — Administered as per standard-of-care.

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug known as LY2963016 as compared to LANTUS® in adults with type 2 diabetes mellitus who are on 2 or more oral antihyperglycemic medications (OAMs).

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM).
* Have been receiving 2 or more OAMs at stable doses for the 12 weeks prior to screening, with or without basal insulin.
* If currently on basal insulin, must be taking LANTUS® QD or NPH or insulin detemir either QD or twice a day for at least 90 days prior to study entry.
* Have an HbA1c ≥7.0% and ≤11.0% if insulin naïve; if previously on basal insulin, then HbA1c ≤11.0%.
* Body mass index (BMI) ≤45 kilograms per meter squared (kg/m^2).
* As determined by the investigator, are capable and willing to do the following:

  * perform self monitored blood glucose (SMBG)
  * complete participant diaries as instructed
  * are receptive to diabetes education
  * comply with required study treatment and study visits

Exclusion Criteria:

* Have been on LANTUS® more than once daily within the previous 30 days.
* Have used any other insulin except the entry insulin [LANTUS®, insulin detemir, or NPH] including commercial (includes any premixed insulins) and investigational insulins within the previous 30 days.
* Have been exposed to a biosimilar insulin glargine within the previous 90 days.
* Have participated in a LY2963016 study.
* Have taken basal plus mealtime insulin (basal bolus therapy) within the last year for greater than 4 continuous weeks.
* Have used any glucagon like peptide (GLP-1) receptor agonists within the previous 90 days.
* Have used pramlintide within the previous 30 days.
* Have excessive insulin resistance at study entry (total insulin dose ≥1.5 units/kg).
* Have more than 1 episode of severe hypoglycemia within 6 months prior to screening.
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the 6 months prior to screening.
* Have known hypersensitivity or allergy to LANTUS® or its excipients.
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy or have received such therapy within 4 weeks immediately preceding screening.
* Have obvious signs or symptoms, or laboratory evidence, of liver disease.
* Have one of the following concomitant diseases: significant cardiac (e.g., congestive heart failure Class III or IV) or gastrointestinal disease (e.g., significant gastroparesis).
* Have a history of renal transplantation or are currently receiving renal dialysis.
* Have a serum creatinine greater than 2.0 milligrams/deciliter (177 micromoles/liter).
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia.
* Participants with active cancer or personal history of cancer within the previous 5 years (with the exception of basal cell carcinoma or carcinoma in situ).
* Have a history or diagnosis of Human Immunodeficiency Virus (HIV) infection.
* Have any other condition (including known drug or alcohol abuse or psychiatric disorder including dementia) that precludes the participant from following and completing the protocol.
* Are pregnant or intend to become pregnant during the course of the study.
* Women who are breastfeeding.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device other than LY2963016, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (10):
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Atlanta Vanguard Medical Associates, Smyrna, Georgia
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Manhattan Medical Research, New York, New York
  - Aventiv Research, Columbus, Ohio
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Advanced Research Institute, South Ogden, Utah
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
- India (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kormangala
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Panjim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Visakhapatnam
- Puerto Rico (2):
  - Manati Center for Clinical Research Inc, Manatí
  - American Telemedicine Center, San Juan
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheboksary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
- South Korea (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ansan-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeju City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Mohan V, Ahn KJ, Cho YM, Sahay RK, Huang CN, Kalra S, Chadha M, Bhattacharya I, Kim SY, Spaepen E. Lilly Insulin Glargine Versus Lantus(R) in Type 2 Diabetes Mellitus Patients: India and East Asia Subpopulation Analyses of the ELEMENT 5 Study. Clin Drug Investig. 2019 Aug;39(8):745-756. doi: 10.1007/s40261-019-00798-1. PMID 31119716
- [Derived] Pollom RK, Ilag LL, Lacaya LB, Morwick TM, Ortiz Carrasquillo R. Lilly Insulin Glargine Versus Lantus(R) in Insulin-Naive and Insulin-Treated Adults with Type 2 Diabetes: A Randomized, Controlled Trial (ELEMENT 5). Diabetes Ther. 2019 Feb;10(1):189-203. doi: 10.1007/s13300-018-0549-3. Epub 2019 Jan 2. PMID 30604091
- See also: Click here for more information about this study: A Study of LY2963016 Compared to LANTUS® in Adult Participants With Type 2 Diabetes Mellitus — http://www.lillytrialguide.com/EN/studies/diabetes/aber

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2963016: Insulin naive participants started on 10 units (U) LY2963016 given subcutaneously (SC) once a day (QD) for 24 weeks. Participants entering the study on LANTUS®, insulin detemir or neutral protamine Hagedorn (NPH) QD were started at the same dose SC. Participants entering on insulin detemir or NPH twice a day (BID) were started at 80% of the total daily dose SC. Participants-driven titration was followed to include the addition of 1 U/day until the fasting blood glucose (FBG) level reaches ≤100 mg/dL (5.6 mmol/L). Participants were allowed to continue oral antihyperglycemic medication (OAM).
- LANTUS®: Insulin naive participants started on 10 U LANTUS® given SC QD for 24 weeks. Participants entering the study on LANTUS®, insulin detemir or NPH QD were started at the same dose SC. Participants entering on insulin detemir or NPH twice a day were started at 80% of the total daily dose SC. Participants-driven titration was followed to include the addition of 1 U/day until the fasting blood glucose (FBG) level reaches ≤100 mg/dL (5.6 mmol/L). Participants were allowed to continue oral antihyperglycemic medication (OAM).
Period: Overall Study
Arm/Group | LY2963016 | LANTUS®
Started | 249 | 244
Received at Least 1 Dose of Study Drug | 249 | 244
Completed | 230 | 225
Not Completed | 19 | 19
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 3 | 4
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2963016 | LANTUS® | Total
Number analyzed (Participants) | 249 | 244 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.82 (8.83) | 56.98 (9.86) | 57.40 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 118 | 236
  Male | 131 | 126 | 257
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 116 | 118 | 234
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 115 | 110 | 225
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 47 | 45 | 92
  Puerto Rico | 29 | 33 | 62
  Turkey | 15 | 10 | 25
  United States | 60 | 57 | 117
  Taiwan | 20 | 22 | 42
  India | 49 | 51 | 100
  Russia | 29 | 26 | 55
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of glycosylated hemoglobin | 8.66 (1.09) | 8.56 (1.02) | 8.61 (1.06)
Sulfonylurea Group [Count of Participants; unit: Participants]
  Yes, did use sulfonylurea | 207 | 207 | 414
  No, did not use sulfonylurea | 42 | 37 | 79
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 11.59 (6.34) | 12.26 (6.45) | 11.92 (6.40)
Time of basal insulin injection [Count of Participants; unit: Participants] — Number of participants who administered a basal insulin injection during the Daytime and Evening/Bedtime.
  Participants
    Daytime | 99 | 96 | 195
    Evening/Bedtime | 150 | 148 | 298

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with baseline of response, treatment (LY2963016, LANTUS), pooled country, basal insulin at entry (yes/no), sulfonylurea (SU) use (yes/no), visit, treatment and visit*treatment in the model.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who received at least 1 dose of study drug and with a Baseline and at least 1 post-Baseline HbA1c measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 226 | 223
Percentage of glycosylated hemoglobin | -1.25 (0.066) | -1.22 (0.067)
Statistical Analysis 1: Comparison: LY2963016 vs LANTUS®; Test type: Non-Inferiority or Equivalence — The primary treatment comparison was to compare LY2963016 versus Lantus at the non-inferiority margin of +0.4%. If the upper limit of the 95% confidence interval on the change from baseline to 24-week HbA1c level for LY2963016 versus Lantus was below +0.4%, then LY2963016 would be declared non-inferior to Lantus; p = 0.693, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.22 to 0.15]

2. Secondary Outcome: Percentage of Participants With HbA1c <7% and ≤6.5%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Endpoint [up to 24 weeks]
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline HbA1c measure; last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 240 | 240
Percentage of participants
  HbA1c- at 24 week endpoint (LOCF) < 7.0% | 35.0 | 38.3
  HbA1c- at 24 week endpoint (LOCF) <= 6.5% | 20.8 | 18.8

3. Secondary Outcome: Change From Baseline in 7-point Self-Monitored Blood Glucose (SMBG) Values
Description: Seven-point SMBG are completed at the following timepoints: Before Morning Meal, 2 Hours After Morning Meal, Before Mid-Day Meal, 2 Hours After Mid-Day Meal, Before Evening Meal, Bed Time and 03:00 AM hours. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline SMBG measure.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 198 | 198
Millimoles per liter (mmol/L)
  24 week- Before Morning Meal | -2.37 (0.083) | -2.69 (0.083)
  24 week- 2 Hours After Morning Meal: number analyzed (Participants) | 187 | 193
  24 week- 2 Hours After Morning Meal | -2.78 (0.161) | -3.00 (0.160)
  24 week-Before Mid-Day Meal: number analyzed (Participants) | 190 | 197
  24 week-Before Mid-Day Meal | -2.14 (0.135) | -2.20 (0.132)
  24 weeks- 2 Hours After Mid-Day Meal: number analyzed (Participants) | 187 | 194
  24 weeks- 2 Hours After Mid-Day Meal | -2.26 (0.158) | -2.42 (0.156)
  24 weeks-Before Evening Meal: number analyzed (Participants) | 190 | 197
  24 weeks-Before Evening Meal | -1.84 (0.156) | -2.25 (0.154)
  24 weeks- Bed Time: number analyzed (Participants) | 189 | 195
  24 weeks- Bed Time | -2.14 (0.157) | -2.40 (0.156)
  24 weeks- 3:00 AM hrs: number analyzed (Participants) | 180 | 189
  24 weeks- 3:00 AM hrs | -2.09 (0.124) | -2.09 (0.122)

4. Secondary Outcome: Intra-Participant Variability in Fasting Blood Glucose (FBG)
Description: Fasting blood glucose (FBG) is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. Intra-Participant FBG variability was calculated based on the standard deviation (SD) of the morning pre-meal BG value. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline fasting blood glucose measure.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 184 | 183
mmol/L | 0.81 (0.049) | 0.79 (0.049)

5. Secondary Outcome: Basal Insulin Dose Units Per Day
Description: Units of Basal Insulin dose taken per day (U/day). Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline Basal Insulin Dose.
Measure: Least Squares Mean (Standard Error); unit: Units per day (U/day)
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 231 | 225
Units per day (U/day) | 49.8 (2.16) | 49.7 (2.17)

6. Secondary Outcome: Basal Insulin Dose Per Body Weight (U/kg/Day)
Description: Basal Insulin dose in units (U) per body weight in kilograms (kg) per day. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline Basal Insulin Dose per Body Weight measure.
Measure: Least Squares Mean (Standard Error); unit: units per kilogram per day (U/kg/day)
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 229 | 225
units per kilogram per day (U/kg/day) | 0.58 (0.024) | 0.61 (0.024)

7. Secondary Outcome: Change From Baseline to 24 Weeks in Body Weight
Description: Change from baseline in body weight. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline body weight measure.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 229 | 225
Kilogram (kg) | 2.3 (0.28) | 1.7 (0.29)

8. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Score
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. Items divided into 5 domains of satisfaction: Inconvenience of Regimen [(IR) 5 items: domain scores range (DSR) 5-35], Lifestyle Flexibility [(LF) 3 items: DSR 3-21], Glycemic Control [(GC) 3 items: DSR 3-21], Hypoglycemic Control [(HC) 5 items: DSR 5-35], Insulin Delivery Device [(IDD) 6 items: DSR 6-42]. All items measured on a 7-point scale: 1 (no bother at all) to 7 (a tremendous bother), with lower scores reflecting better outcomes. ITSQ Total Overall Raw Scores range from 22-154. Both raw domain and overall scores are transformed on a scale of 0-100, where transformed score=100*[(7-mean raw score)/6]. Higher scores indicate better treatment satisfaction. LS means was determined by MMRM with baseline of response, baseline HbA1c, country, sulfonylurea use, basal insulin status at study entry, visit, treatment and visit*treatment in the model.
Time Frame: Week 4 and Week 24
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline ITSQ measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 234 | 235
units on a scale
  IR-Week 4 | 85.79 (1.32) | 84.92 (1.33)
  IR-Week 24: number analyzed (Participants) | 230 | 225
  IR-Week 24 | 84.75 (1.26) | 84.91 (1.28)
  LF-Week 4 | 71.43 (1.87) | 69.11 (1.89)
  LF-Week 24: number analyzed (Participants) | 230 | 225
  LF-Week 24 | 72.44 (1.77) | 70.87 (1.80)
  HC-Week 4 | 77.82 (1.50) | 76.98 (1.52)
  HC-Week 24: number analyzed (Participants) | 230 | 225
  HC-Week 24 | 76.18 (1.46) | 76.52 (1.48)
  GC-Week 4 | 79.24 (1.45) | 78.87 (1.46)
  GC-Week 24: number analyzed (Participants) | 230 | 224
  GC-Week 24 | 82.14 (1.36) | 81.30 (1.38)
  IDD-Week 4: number analyzed (Participants) | 233 | 235
  IDD-Week 4 | 82.21 (1.23) | 82.37 (1.25)
  IDD-Week 24: number analyzed (Participants) | 230 | 225
  IDD-Week 24 | 82.12 (1.29) | 82.01 (1.31)
  ITSQ Overall Total-Week 4 | 80.15 (1.12) | 79.40 (1.13)
  ITSQ Overall Total-Week 24: number analyzed (Participants) | 230 | 225
  ITSQ Overall Total-Week 24 | 80.01 (1.13) | 79.76 (1.14)

9. Secondary Outcome: Percentage of Participants With Detectable Anti-Drug Antibodies to LY2963016 or LANTUS®
Description: The percentage of participants with detected insulin antibodies were summarized as counts and percentages at baseline, at each visit, at the 24-week endpoint (LOCF), and overall for the 24-week treatment period.
Time Frame: Endpoint [up to 24 weeks]
Population: All randomized participants who received at least 1 dose of study drug and with a Baseline and at least 1 post-Baseline with detectable anti-drug antibodies; last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 234 | 239
Percentage of participants | 14.5 | 17.2

10. Secondary Outcome: Rate of Hypoglycemic Events Adjusted Per 1 Year
Description: The rate of hypoglycemic events were analyzed at baseline, titration, maintenance, and overall study periods and at endpoint using the Wilcoxon test. In addition, a negative binomial model was used as a sensitivity analysis. A hypoglycemic event is defined as any time a participant has a blood glucose (BG) level of ≤70 milligrams per deciliter (mg/dL) even if the event was not associated with signs, symptoms, or treatment consistent with current guidelines (American Diabetes Association 2005). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking. Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrates, glucagons, or other resuscitative actions. Severe Hypoglycemic events may or may not have a reported BG ≤70 mg/dL. These events may be associated with sufficient neuroglycopenia to induce seizure or coma.
Time Frame: Baseline through Endpoint [up to 24 weeks]
Population: All randomized participants who received at 1 dose of study drug with Baseline at least 1 post-Baseline hypoglycemic event; last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Hypoglycemic events per 1 year
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 246 | 243
Hypoglycemic events per 1 year
  Total Hypoglycemia with BG ≤70 mg/dL | 16.95 (23.444) | 23.37 (35.809)
  Severe Hypoglycemia | 0.00 (0.00) | 0.00 (0.02)
  Nocturnal Hypoglycemia with BG ≤70 mg/dL | 6.64 (11.650) | 7.94 (17.882)

11. Secondary Outcome: Percentage of Participants With Hypoglycemic Events
Description: The percentage of participants (with at least 1 hypoglycemic event (total, severe, nocturnal, and others) or incidence during the study was analyzed using Fisher's exact test. A hypoglycemic event is defined as any time a participant has a blood glucose (BG) level of ≤70 milligrams per deciliter (mg/dL) even if the event was not associated with signs, symptoms, or treatment consistent with current guidelines (American Diabetes Association 2005). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking. Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrates, glucagons, or other resuscitative actions. Severe Hypoglycemic events may or may not have a reported BG ≤70 mg/dL. These events may be associated with sufficient neuroglycopenia to induce seizure or coma.
Time Frame: Endpoint [up to 24 weeks]
Population: All randomized participants who had a post-baseline measurement for Hypoglycemic Events; last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | LY2963016 | LANTUS®
Number analyzed (Participants) | 249 | 244
Percentage of participants
  Total hypoglycemia with BG ≤70 mg/dL | 68.7 | 69.1
  Severe hypoglycemia | 0 | 0.8
  Nocturnal hypoglycemia with BG ≤70 mg/dL | 49.6 | 46.1
  Non-nocturnal hypoglycemia with BG ≤70 mg/dL | 59.4 | 63.0

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: All the randomized participants who received at least one dose of the study drug.
Arm/Group | LY2963016 | LANTUS®
Serious Adverse Events (participants affected / at risk) | 10/249 | 12/244
Other Adverse Events (participants affected / at risk) | 75/249 | 87/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=249) | LANTUS® (N=244)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=249) | LANTUS® (N=244)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Fatigue (General disorders) | 2 (2) | 3 (3)
Injection site pain (General disorders) | 2 (2) | 7 (11)
Pyrexia (General disorders) | 3 (3) | 4 (5)
Bronchitis (Infections and infestations) | 3 (3) | 3 (4)
Nasopharyngitis (Infections and infestations) | 18 (23) | 24 (26)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 9 (10)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Viral infection (Infections and infestations) | 3 (3) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Weight increased (Investigations) | 8 (9) | 4 (4)
Abnormal weight gain (Metabolism and nutrition disorders) | 7 (9) | 5 (7)
Vitamin d deficiency (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Hypertension (Vascular disorders) | 3 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days